CLINICAL TRIAL: NCT03272698
Title: A Prospective Randomized Controlled Trial of Electroconvulsive Therapy with Ketamine Anesthesia (Standard Therapy) and High Intensity Ketamine with Electroconvulsive Therapy Rescue for Treatment-Resistant Depression - EAST HIKER Trial
Brief Title: ECT with Ketamine Anesthesia Vs High Intensity Ketamine with ECT Rescue for Treatment-Resistant Depression
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Royal University Hospital Foundation (Other)
Responsible Party: Principal Investigator, Jonathan Gamble, M.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2017-08-28; First posted 2017-09-05 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Treatment Resistant Depression; Ketamine
Keywords: ketamine; treatment-resistant depression; electroconvulsive therapy
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Patients in the EAST arm will receive eight ECT sessions (on a bi/triweekly schedule, weekdays only) with ketamine-based general anesthetic (ketamine 0.75 mg/kg, remifentanil 1 mcg/kg, and succinylcholine 0.75 mg/kg for safety. Patients in the HIKER arm will receive a single dose of ketamine 0.50 mg/kg, on 8 successive weekdays. Since ketamine without ECT is not the standard of care for TRD, patients in the HIKER arm who do not achieve a 25% reduction in the Montgomery-Asberg Depression Rating Scale (MADRS) after the third treatment will be deemed non-responsive to ketamine and switched to a standard 8 treatment course of ECT with ketamine-based GA as described in the EAST arm - this will be called rescue ECT. The attending psychiatrist may discontinue therapy for either arm if the patient achieves remission or treatment is ineffective based on clinical judgment.
Who Masked: Investigator
Masking Description: Patients will be randomized to either the HIKER or EAST arms, but due to the different frequencies of treatment, patient and physician blinding will not be possible. Outcome assessor will also not be blinded. As patients were not blinded, they could easily divulge their treatment allocation. The outcome assessor can also deduce treatment allocation from communications with nursing staff or study personnel. However, the follow up assessment at 30 days post-final treatment will be performed by a different study team member who will remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine (HIKER) (Experimental): Patients in the HIKER arm will receive a single dose of ketamine 0.50 mg/kg, which is enough to achieve a full anaesthetic effect (i.e., unconsciousness mimicking the GA regimen above), on 8 successive weekdays.
  Interventions: Drug: Ketamine
- Ketamine-ECT (EAST) (Active Comparator): Patients in the EAST arm will initially receive intravenous ketamine 0.75 mg/kg, remifentanil 1 mcg/kg (to reduce discomfort), and succinylcholine 0.75 mg/kg (for safety). Based on patients' anaesthetic response, the attending anaesthesiologist is given the freedom to vary the dose of remifentanil and succinylcholine as well as administer propofol to achieve safe and acceptable anaesthetic conditions. As per the Saskatoon Health Region's care standard, patients in the EAST arm will receive eight ECT sessions (on a bi/triweekly schedule) delivered by the attending psychiatrist with either unilateral or bilateral electrode placement and monitoring of seizure threshold by the half-age method.
  Interventions: Drug: Ketamine; Procedure: ECT

INTERVENTIONS:
Drug: Ketamine — IV Ketamine 0.50 mg/kg
  Other Names: Ketalar
Procedure: ECT — ECT with unilateral or bilateral electrode placement and monitoring of seizure threshold by the half-age method
  Arms: Ketamine-ECT (EAST)

SUMMARY:
To determine if an high intensity ketamine with ECT rescue (HIKER) approach for treatment resistant depression will: 1) reduce patient suffering by hastening disease remission, 2) have fewer side effects, 3) reduce the need for ECT, and 4) be preferred by most patients. Half of participants will be randomized to the HIKER arm and receive high intensity ketamine treatment for eight consecutive days, and the other half will be assigned to the ECT with ketamine anesthesia (EAST) arm and receive 8 ECT treatments (2-3 treatment/week)

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common psychiatric illness that will affect at least 15% of the population. The burden of MDD is staggering, considered by the World Health Organization to be the leading cause of disability in developed countries for people aged 15-44.

Oral antidepressant therapy for MDD is notoriously ineffective. At least 3 weeks of treatment is usually required to achieve response rates that rarely exceed 40% (only 10% better than placebo); furthermore, treatment can be complicated by serious side effects serious (e.g. falls, weight gain) including increased suicidality. Up to 15% of patients will eventually be diagnosed as having treatment-resistant depressions (TRD), defined as the failure to respond to at least two antidepressants from different pharmacologic classes after adequate treatment duration at therapeutic dosages. The gold standard therapy for TRD is electroconvulsive therapy (ECT) with general anaesthesia (GA), which produces rapid antidepressant effects after only a few sessions. Propofol is the traditional anaesthetic agent used in GA for ECT, although recently this research group showed that ECT with ketamine as the primary anaesthetic produced faster depression remission compared to ECT with propofol.

Despite its efficacy, ECT is associated with considerable problems. More than 10% of patients will experience amnesia and confusion, which can persist for weeks. These cognitive side effects limit the frequency of ECT treatments to two or three times per week. There is also a risk of rare but devastating cardiorespiratory adverse events, at least part of which can be attributed to the need to induce chemical paralysis (for safety) and administer opioids (for pain control) during ECT with GA. Lastly, ECT requires specialized psychiatric expertise, dedicated resources, specially trained nurses, and an anaesthesiologist - requirements that are both costly and not readily available in many settings.

In contrast to ECT, daily short-acting anaesthesia, including ketamine, is well tolerated. A recent study found that only three treatments of intravenous ketamine produced a greater early improvement in depression scores compared to ECT under non-ketamine-based GA. This suggests a possibility of achieving early disease remission in TRD with ketamine-only infusions while avoiding the safety risks and treatment delays associated with ECT under GA.

The efficacy, feasibility, and improved side-effect profile of frequent successive ketamine treatments suggest it may be the preferred treatment for TRD compared to ECT with ketamine-based GA. There may, however, be a small subgroup of TRD patients who do not respond to ketamine alone and require ECT, although with a daily treatment regimen, ketamine non-responders could be quickly identified and given a standard course of ECT. The researchers propose that a treatment protocol of daily High Intensity Ketamine with ECT Rescue (HIKER) will be superior to ECT Therapy with ketamine anesthesia standard therapy (EAST) in facilitating early disease remission, while at the same time yielding similar overall remission rates by allowing ketamine non-responders to be quickly identified and given ECT.

ELIGIBILITY:
Inclusion Criteria:

* Montgomery Asberg Depression Rating Scale (MADRS) score of greater than 20) planned for ECT therapy.
* Subjects must meet clinical criteria for TRD defined as failure to respond to at least 2 standard-of-care drug therapies of adequate treatment duration.

Exclusion Criteria:

* Subjects will be ineligible if they cannot provide informed consent
* American Society of Anesthesiology physical status score of four or greater
* Implanted medical device with electronic parts (e.g. pacemaker, defibrillator, intrathecal pump, spinal cord stimulator, deep brain stimulator)
* Schizoaffective disorder
* Women of child-bearing potential will be asked to undergo a commercial urine pregnancy screening test. Those who refuse or screen positive will be excluded.
* Allergic to any of the study drugs or their carrier components
* Any serious physical condition prior to randomization deemed by the attending psychiatrist or consulting anesthetist to be a contraindication to ECT such as cardiovascular disease (including untreated hypertension), respiratory disease, cerebrovascular disease, intracranial hypertension (including glaucoma), or seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of treatments required to reach disease remission | From date of randomization until the date of disease remission or after 8 treatments, assessed up to 4 weeks
  The primary outcome is number of treatments required to reach disease remission, as defined by a reduction of MADRS score to under 10

SECONDARY OUTCOMES:
Rate of rescue ECT in the HIKER arm | From date of randomization up to 6 days
  Percent of patients in the HIKER arm who do not achieve a 25% reduction in the Montgomery-Asberg Depression Rating Scale (MADRS) after the third treatment.
Suicidal ideation | From date of randomization until the date of disease remission or after 8 treatments and at 30 days following last treatment, assessed up to 8 weeks
  Suicidal ideation as measured by the Columbia Suicide Severity Rating Scale
Cognitive Impairment | MMSE will be assessed at baseline, final treatment, and 30 day post-treatment follow-up
  Cognitive Impairment as measured by Mini-Mental State Exam (MMSE)
Self- and clinician rated improvement | From date of randomization until the date of disease remission or after 8 treatments and at 30 days following last treatment, assessed up to 8 weeks
  Patients will rate their condition on the patient-rated clinical global impression - improvement scale (PGI-I)
Patient satisfaction with treatment | From date of randomization until the date of disease remission or after 8 treatments and at 30 days following last treatment, assessed up to 8 weeks
  Satisfaction with treatment will be assessed by the 2-item treatment satisfaction questionnaire for medication-version II (TSQM-GS-II).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gamble, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Mathers C, Fat DM, Boerma JT. The global burden of disease: 2004 update: World Health Organization; 2008.
- [Background] Kirsch I, Deacon BJ, Huedo-Medina TB, Scoboria A, Moore TJ, Johnson BT. Initial severity and antidepressant benefits: a meta-analysis of data submitted to the Food and Drug Administration. PLoS Med. 2008 Feb;5(2):e45. doi: 10.1371/journal.pmed.0050045. PMID 18303940
- [Background] Skolnick P, Layer RT, Popik P, Nowak G, Paul IA, Trullas R. Adaptation of N-methyl-D-aspartate (NMDA) receptors following antidepressant treatment: implications for the pharmacotherapy of depression. Pharmacopsychiatry. 1996 Jan;29(1):23-6. doi: 10.1055/s-2007-979537. PMID 8852530
- [Background] Berlim MT, Turecki G. Definition, assessment, and staging of treatment-resistant refractory major depression: a review of current concepts and methods. Can J Psychiatry. 2007 Jan;52(1):46-54. doi: 10.1177/070674370705200108. PMID 17444078
- [Background] Fink M. Is Catatonia a Primary Indication for ECT? Convuls Ther. 1990;6(1):1-4. No abstract available. PMID 11941041
- [Background] Bundy BD, Hewer W, Andres FJ, Gass P, Sartorius A. Influence of anesthetic drugs and concurrent psychiatric medication on seizure adequacy during electroconvulsive therapy. J Clin Psychiatry. 2010 Jun;71(6):775-7. doi: 10.4088/JCP.08m04971gre. Epub 2009 Dec 29. PMID 20051218
- [Background] Comparing Ketamine and Propofol Anesthesia for Electroconvulsive Therapy [database on the Internet]. 2013 [cited 2017 Jan 1]
- [Background] Datto CJ. Side effects of electroconvulsive therapy. Depress Anxiety. 2000;12(3):130-4. doi: 10.1002/1520-6394(2000)12:33.0.CO;2-C. PMID 11126187
- [Background] Ghasemi M, Kazemi MH, Yoosefi A, Ghasemi A, Paragomi P, Amini H, Afzali MH. Rapid antidepressant effects of repeated doses of ketamine compared with electroconvulsive therapy in hospitalized patients with major depressive disorder. Psychiatry Res. 2014 Feb 28;215(2):355-61. doi: 10.1016/j.psychres.2013.12.008. Epub 2013 Dec 13. PMID 24374115
- [Background] Metriyakool K. Methohexital as alternative to propofol for intravenous anesthesia in children undergoing daily radiation treatment: a case report. Anesthesiology. 1998 Mar;88(3):821-2. doi: 10.1097/00000542-199803000-00035. No abstract available. PMID 9523828
- [Background] Irwin SA, Iglewicz A, Nelesen RA, Lo JY, Carr CH, Romero SD, Lloyd LS. Daily oral ketamine for the treatment of depression and anxiety in patients receiving hospice care: a 28-day open-label proof-of-concept trial. J Palliat Med. 2013 Aug;16(8):958-65. doi: 10.1089/jpm.2012.0617. Epub 2013 Jun 27. PMID 23805864
- [Background] Diamond PR, Farmery AD, Atkinson S, Haldar J, Williams N, Cowen PJ, Geddes JR, McShane R. Ketamine infusions for treatment resistant depression: a series of 28 patients treated weekly or twice weekly in an ECT clinic. J Psychopharmacol. 2014 Jun;28(6):536-44. doi: 10.1177/0269881114527361. Epub 2014 Apr 3. PMID 24699062
- [Background] Rush AJ, Blacker D. Handbook of psychiatric measures: American Psychiatric Pub; 2008
- [Background] Gipson PY, Agarwala P, Opperman KJ, Horwitz A, King CA. Columbia-suicide severity rating scale: predictive validity with adolescent psychiatric emergency patients. Pediatr Emerg Care. 2015 Feb;31(2):88-94. doi: 10.1097/PEC.0000000000000225. PMID 25285389
- [Background] Atkinson MJ, Kumar R, Cappelleri JC, Hass SL. Hierarchical construct validity of the treatment satisfaction questionnaire for medication (TSQM version II) among outpatient pharmacy consumers. Value Health. 2005 Nov-Dec;8 Suppl 1:S9-S24. doi: 10.1111/j.1524-4733.2005.00066.x. PMID 16336491
- [Background] Guy W. Clinical global impression scale. The ECDEU Assessment Manual for Psychopharmacology-Revised Volume DHEW Publ No ADM. 1976;76(338):218-22